CLINICAL TRIAL: NCT01359683
Title: Heart Rate Variability Changes During Cardiac Surgery And The Incidence Of Post-Operative Cardiac Arrhythmias
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University College of Medicine (Other)
Responsible Party: Sponsor
Organization: Drexel University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17028
Record Dates: First submitted 2008-04-07; First posted 2011-05-25 (Estimated); Last update posted 2013-06-14 (Estimated); Status verified 2008-04

CONDITIONS: Cardiac Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Other): This is a prospective observational study. 100 patients in one arm scheduled for cardiac surgery will be enrolled. ECG tracings will be obtained when subject is at rest, in supine position, before induction of anesthesia (within 24 hours prior to induction), after induction of general anesthesia, right before emergence from anesthesia (or before transportation to the ICU if the subject remains intubated), and within 24 hours post-operatively; additional ECG readings may be obtained during the surgery if deemed necessary.
  Interventions: Device: Dataq Instruments DI-158

INTERVENTIONS:
Device: Dataq Instruments DI-158 — Data Acquisition Device (connects to room instrumentation)

SUMMARY:
The purpose of this study is to investigate non-linear heart rate variability indexes as predictors of the incidence of cardiac arrhythmias in patients undergoing cardiac surgery, including coronary artery bypass graft (CABG) and valvular surgery.

ELIGIBILITY:
Inclusion Criteria:

* All patients who will have cardiac surgery
* The patient must be mentally able and willing to participate in the study
* Male or female patients over the age of 18

Exclusion Criteria:

* Patients with major renal, hepatic, respiratory, or cerebral dysfunction
* Patients with atrial fibrillation or other forms of sinus node dysfunction
* Patients requiring continuous artificial pacing
* Patients with significant congenital heart disease with or without arrhythmias
* Patients on Intra-Aortic Balloon Pump
* Patients experiencing cardiac emergencies or undergoing cardiac salvage operations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-09; Primary Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Investigate non-linear heart rate variability (HRV) indexes as predictors of the incidence of cardiac arrhythmias in patients undergoing cardiac surgery, including coronary artery bypass graft (CABG) and valvular surgery. | Sept 07 - Sept 08

SECONDARY OUTCOMES:
Registration of HRV changes during cardiac surgery, and comparison HRV pre-operatively, post anesthesia induction, on emergence from anesthesia and postoperatively. | Sept 07 - Sept 08

CONTACTS AND LOCATIONS:
Locations (1):
- Hahnemann University Hospital, Philadelphia, Pennsylvania, United States